CLINICAL TRIAL: NCT05334082
Title: Effects of the FIFA 11+ on Physical Performance and Injury Prevention in Female Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, MARIO ALEXANDRE GONÇALVES LOPES, Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIFA11+FemaleFutsal
Record Dates: First submitted 2022-03-22; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Injuries; Flexibility; Balance
Keywords: Velocity; Epidemiology; Warm-up; Pliometric; Injury burden
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Experimental, randomized, controlled and multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ Group (Experimental): Teams will replace regular warm-up with the intervention protocol - FIFA11+ injury prevention program - during training sessions
  Interventions: Other: FIFA 11+
- Control Group (No Intervention): Teams will maintain regular warm-up during training sessions

INTERVENTIONS:
Other: FIFA 11+ — 15 progressive exercise drills for training preparation (warm-up)
  Other Names: Injury prevention program
  Arms: FIFA 11+ Group

SUMMARY:
The FIFA 11 + is an injury prevention that has shown to improve physical performance and prevent injuries in male futsal players, however, this injury prevention program has not been tested in female futsal players.

The investigators aim to test the effects of the FIFA 11 + program on physical performance and injury prevention in female futsal players.

DETAILED DESCRIPTION:
According to the FIFA Medical Assessment and Research Center (F-MARC), consistent implementation of the "11+" program can lead to a 30-50% reduction in injuries. As the practice of soccer implies risk of injury, as well as F-MARC, considers that during training you should also include exercises to reduce the risk of injury. This warm-up program is intended to replace the traditional pre-workout warm-up. According to F-MARC, the key elements in injury prevention programs for footballers are core strength, neuromuscular control and balance, eccentric hamstring training, plyometrics and agility. The FIFA 11 has shown to improve physical performance and prevent injuries in male futsal players, however, this injury prevention program has not been tested in female futsal players.

With an experimental, randomized, controlled and multicenter study, the investigators intend to verify if the FIFA "11+" reduces injuries and produces changes in proprioception, static and dynamic balance, muscle strength, plyometric and agility results different from traditional warm-up/training programs used in futsal in 10 weeks.

The study will be carried out during the 2021/22 season, in the first division of the senior female national championships with a sample of 60 athletes. It is intended to implement a rigorous methodological process that allows solving the methodological problems of previous studies. The investigators will also characterize the injury profile of female futsal players in Portugal.

The present study intends to include all injuries sustained by players throughout the abovementioned time period. Injuries will be categorized according to type, location, mechanism of injury (traumatic or overuse), whether the injury was a recurrence onset, severity and if it was during training or match. Injury definition and classification will be set in accordance to the consensus agreement of injury definitions: slight (0 days), minimal (1-3 days), mild (4-7 days), moderate (8-28 days), severe (>28 days) and career ending. Injury-related data will follow the Consensus statement on injury definitions.

Anthropometric data will include, sex, age, height; weight, body mass index (BMI).Technical data will include lower limb dominance; players' playing position (keeper, lastman, winger, pivot and wing-pivot) age of initiation of futsal practice.

All analyses will be conducted on SPSS version 24.0 (SPSS Inc., Chicago, IL, USA). Normality of data distribution will be tested with the Shapiro-Wilk test. Descriptive statistics will be used to calculate the mean and standard deviation (SD). Injury incidence rates (number of injuries/1000 player-hours) will be calculated for all selected groups.

Dispersion in these variables was expressed as typical deviation and/or maximum and minimum values. Normality was studied using the Kolmogorov-Smirnoff test. Qualitative variables were expressed as absolute frequency and percentage. Quantitative variables were contrasted using the Kruskal-Wallis test for independent samples. Qualitative variables were analyzed using contingency tables and their statistical significance using Pearson's 12 test. All hypothesis contrasts performed were bilateral, taking a value of p<0.05 as statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Futsal players enrolled in the Official Futsal Championship of the Portuguese Football Federation;
* Attendance of at least 50% of training sessions;

Exclusion criteria:

- Clinical diagnosis of cancer, arthritis, heart disease, pulmonary disease, neurological disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Injuries sustained | 6 months
  injuries sustained during the study period
Characteristics of the injury sustained | 6 months
  Trauma/overuse, body location, ligament/muscle injury
Recovery time | 6 months
  days of recovery until return-to-play
Training exposure | 6 months
  minutes of training
Match exposure | 6 months
  minutes of match play
Number of FIFA 11+ sessions | 6 months
  number of FIFA 11+ sessions attended during the study period

SECONDARY OUTCOMES:
Speed | 10 weeks
  30m sprint (sec)
Jump performance | 10 weeks
  single and double leg hop test (distance jumped - cm)
Agility | 10 weeks
  T-Agility test (sec)
Flexibility | 10 weeks
  sit-and-reach test (cm)
Dynamic balance | 10 weeks
  Y-balance test (%): lower lim reach distance (cm) normalized to the lenght of the lower limb (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde da Universidade de Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
All collected IPD, all IPD that underlie results in a publication.